CLINICAL TRIAL: NCT04956562
Title: Effect of Inactivated COVID-19 Vaccine, Sinovac on Survival in Intensive Care Unit
Brief Title: Effect of Sinovac on Survival in Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Sisli Hamidiye Etfal Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Sultan Acar Sevinç, consultant doctor, Sisli Hamidiye Etfal Training and Research Hospital
Other Study IDs: 1903
Record Dates: First submitted 2021-06-30; First posted 2021-07-09 (Actual); Last update posted 2021-07-09 (Actual); Status verified 2021-06

CONDITIONS: Survival; Intensive Care Unit
Keywords: covid-19 vaccine; sinovac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Vaccinated with sinovac: Vaccinated COVID-19 patients over 65 years consisted the study group
- Unvaccinated: Unvaccinated patients over 65 years composed the control group

SUMMARY:
Effect of Inactivated COVID-19 Vaccine (Sinovac) on survival in intensive care unit, Single Center Experience

DETAILED DESCRIPTION:
Turkey has started vaccinate healthcare professionals at 13 January 2021 by Sinovac vaccine and declared a step by step inclusion schedule The primary aim of the study is to compare clinical, laboratory and survival data of COVID-19 patients who were vaccinated at least 14 days before enrollment to the study with COVID-19 patients not vaccinated although they would have. The secondary aim is to compare age of enrolled patients to ICU due to SARS-CoV-2 infection with patients admitted to ICU before start of vaccination program.

ELIGIBILITY:
Inclusion Criteria:

* Patients with covid 19 over the age of 65 who were admitted to the intensive care unit between 1 April 2021 and 15 May 2021

Exclusion Criteria:

* admissions to ICU due to reasons other than COVID-19, age younger than 65, continued admission at the end of enrolment date,

Min Age: 65 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients admitted to our institution's intensive care unit (ICU) between 01 April 2021 and 15 May 2021 was enrolled to the study. Exclusion criteria was admissions to ICU due to reasons other than COVID-19, age younger than 18, continued admission at the end of enrolment date.
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-05-15 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
survival data | 30 days
  If the patient dies, we have reached an outcome

CONTACTS AND LOCATIONS:
Locations (1):
- Sisli Hamidiye Etfal Research and Training Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Sevinc SA, Metin S, Basi NB, Ling J, Cinar AS, Oba S. Effectiveness of inactivated SARS-CoV-2 vaccine (CoronaVac) on intensive care unit survival. Epidemiol Infect. 2022 Feb 9;150:e35. doi: 10.1017/S0950268822000267. PMID 35135644